CLINICAL TRIAL: NCT03432507
Title: The Association Between Proinflammatory Cytokines, Microbial Infection and Clinical Manifestation in Sciatica Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Eisenberg Elon MD, Elon Eisenberg MD Professor of Neurology and Pain Medicine Head, Pain Research Unit Institute of Pain Medicine Rambam Health Care Campus, Rambam Health Care Campus
Other Study IDs: 0477-17
Record Dates: First submitted 2018-01-31; First posted 2018-02-14 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — dissected intra-vertebral discs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- disc herniation: patients suffering from disc herniation
  Interventions: Other: PCR
- spinal stenosis: patients suffering from spinal stenosis
  Interventions: Other: PCR

INTERVENTIONS:
Other: PCR — PCR for proinflammatory cytokines (IL-1b, IL-6, IL-8, IL-17, TNF-a, INF-g) and bacteria

SUMMARY:
All patients scheduled for lumbar spine surgery due to discogenic low back pain and/or sciatica, will be screened by the principal investigator for presence of inclusion/exclusion criteria. Their baseline neurological function before surgery will be assessed and recorded for recruitment into one of the three study groups. MRI scans will be assessed for the calculation of disc protrusion size. Experimental sensory and pain assessments and questionnaires will be performed at list 24 hours before surgery. Blood sample for pro-inflammatory mediator will be obtained at the same time as the experimental sensory and pain tests. Pre-operative pain and MPQ will be assessed pre-operatively (back and leg pain separately), and again on day 30 after surgery. Blood tests for ESR, CRP will be drawn before surgery, during the surgery, and on 30 after surgery. During surgery, intervertebral disc material will be harvested and divided into 4 specimens for culture and inflammatory mediator analysis. Repeat neurological assessment will be performed 30 after surgery.

DETAILED DESCRIPTION:
The clinical manifestation of disc degeneration and/or disc herniation can be low back pain and/or sciatica. The patterns of sensory and motor signs and symptoms that develop after neuropathy vary between individual patients with disc degeneration and/or disc herniation. The expression of these sensory signs (hyperalgesia, allodynia, and sensory loss), which we call the individual somatosensory profile, reflects pathophysiological mechanisms in damaged and surviving afferent nerve fibers such as conduction block, ectopic impulse generation, peripheral sensitization, and central sensitization. In addition, studies have been conducted in search of a microbial origin responsible for the observed inflammatory reaction in discogenic low back pain and sciatica. However, the studies tested mixed cohorts of patients in terms of clinical symptoms (low back pain alone, sciatica, both), length of symptoms (acute and chronic), and tissue cultured (disc, bone). We hypothesize that the possible infectious etiology of the observed inflammatory reaction seen in acute disc herniation and sciatica may be different from that of chronic low back pain due to disc degeneration.

We further suspect that the immununogenicity of an acute disc herniation causing neurological deficit may be different from a similar disc herniation not causing a deficit, and still different from chronic degenerated discs without herniation or neurological deficit. Despite the frequent occurrence of low back pain and sciatica in the general population their underling mechanisms are poorly understood.

Aims and hypotheses of study

(1) To test the differences in disc microbial cultures and in levels of disc and blood cytokines, between patients suffering disc degeneration / herniation and spinal stenosis (controls), and (2) to assess the relationship between clinical manifestations and sensory profiles of these patients and levels of cytokines found in disc tissue and blood.

Ouer hypotheses are: (1) patients suffering from disc degeneration / herniation or spinal stenosis will differ in microbial culture and cytokines levels, with higher levels of positive microbial disc culture and cytokines in the disc herniation group, (2) proinflamtory cytokines levels will correlate with hyperalgesic (rather than hypoalgesic) sensory profiles.

Methods

200 adult subjects suffering from radicular pain duo to disc degeneration / herniation or spinal stenosis will be recruited from the orthopedic clinic at the Rambam Health Care Campus.

Experimental sensory and pain assessments will include a set of non-painful and pain evoked tests which assess sensory integrity and pain perception to thermal (heat and cold) and mechanical (vibration fork, pressure algometer and Von Frey Filaments) stimulation and an assessment of the pain modulation processes: (1) conditioned pain modulation (CPM)- a phenomenon whereby the response to a given noxious test stimulus is attenuated by another conditioning noxious stimulus which is simultaneously administered in a remote area of the body; (2) temporal summation (TS)- the experimental equivalent of 'windup. The tests will be performed over the skin of the painful area (back and leg) and over the same areas of the non-painful contralateral side. Clinical pain assessments will be based on the evaluation of pain intensity on a daily pain diary as well as on a pain questionnaire (Short-Form McGill Pain Questionnaire (SF-MPQ)); Thermal detection and pain thresholds and the number of paradoxical heat sensations The thermal tests will be performed using the TSA II (MEDOC, Israel). Cold and warm detection thresholds will be measured first (CDT, WDT). In addition, subjects will be asked about paradoxical heat sensations (PHS) during the thermal sensory limen (TSL) procedure of alternating warm and cold stimuli. Then cold pain and heat pain thresholds will be determined (CPT, HPT). The mean threshold temperature of three consecutive measurements will be calculated. All thresholds will be obtained with ramped stimuli (1°C/s) that will be terminated when the subject presses a button. The baseline temperature will be 32°C and the contact area of the thermode will be 3x3 cm2. Cut-off temperatures will be 0°C and 50°C

Mechanical detection and pain threshold The mechanical detection threshold (MDT) will be measured with a standardized set of von Frey hairs (Optihair2-Set, Marstock Nervtest, Germany) that exert forces upon bending between 0.25 and 512 mN (1-2s contact time). The contact area of the von Frey hairs with the skin will be of uniform size and shape (rounded tip, 0.5 mm in diameter) to avoid sharp edges that would facilitate nociceptor activation. Using the ''method of limits'', five threshold determinations will be made, each with a series of ascending and descending stimulus intensities. The final threshold will be the geometric mean of these five series.

The mechanical pain threshold (MPT) will be measured using a standardized set of von Frey hairs. The stimulators will be applied at a rate of 2s on, 2s off in an ascending order until the first percept of sharpness will be reached. The final threshold will be the geometric mean of five series of ascending and descending stimuli. This test will be designed to detect pinprick hypoalgesia.

Stimulus/response-functions: mechanical pain sensitivity for pinprick stimuli and dynamic mechanical allodynia Mechanical pain sensitivity (MPS) will be assessed using the von Frey hair with the strongest force (512 mN). Subjects will be asked to give a pain rating for 35 stimulus on a '0-100' numerical rating scale ('0' indicating ''no pain'', and '100' indicating ''most intense pain imaginable'').

Dynamic mechanical allodynia (ALL) will be assessed using a set of three light tactile stimulators as moving innocuous stimuli: Cotton wisp exerting a force of 3 mN, a cotton wool tip fixed to an elastic strip exerting a force of 100 mN, and a standardized brush exerting a force of 200-400 mN. The tactile stimuli will be applied with a single stroke of approximately 2 cm in length over the skin. Fifteen stimuli will be given (five per stimulus type). All stimuli will be applied with a 10s inter-stimulus interval - well below the critical frequency for wind-up. Mechanical pain sensitivity will be calculated as the geometric mean of all numerical ratings for pinprick stimuli. Dynamic mechanical allodynia will be calculated as the geometric mean (compound measure) of all numerical ratings across all three different types of light touch stimulators.

Wind-up ratio representing the perceptual correlate of temporal pain summation In this test, the perceived intensity of a single pinprick (256 mN) will be compared with that of a series of 10 repetitive pinprick stimuli of the same physical intensity (1/s applied within an area of 1 cm2). The subject will be asked to give a pain rating representing the single stimulus, and the estimated mean over the whole series of 10 stimuli using a '0-100' numerical rating scale. The whole procedure will be repeated five times. Wind-up ratio (WUR) will be calculated as the ratio: mean rating of the five series divided by the mean rating of the five single stimuli.

Vibration detection threshold The vibration detection threshold (VDT) represents the only disappearance threshold within the proposed QST battery. This test will be performed with a Rydel-Seiffer grade tuning fork (64 Hz, 8/8 scale) that will be placed over a bony prominence (lateral or medial malleolus) and left there until the subject could not feel vibration any more. Vibration detection threshold will be determined as a disappearance threshold with three stimulus repetitions.

Pressure pain threshold (PPT) The final test in the protocol will be performed over muscle in the painful limb with a pressure gauge device (FDN200, Wagner Instruments, USA) with a probe area of 1 cm2 (probe diameter of 1.1 cm) that exerts forces up to 20 kg/cm2. The pressure pain threshold will be determined with three series of ascending stimulus intensities, each applied as a slowly increasing ramp of 0.5 kg/cm2 s.

Temporal summation of heat pain Noxious heat stimuli will be given to the painful site. The tonic heat pain (THP) stimulation will be applied using the 3 X 3 cm Peltier based computerized thermal stimulator (TSA, Medoc Ltd, Ramat Yishai, Israel). The baseline temperature will be 32ºC and increase at a rate of 2ºC/sec up to a destination temperature of 46.5ºC and will last for 2 minutes. Participants, unaware of the temperature, will be instructed to verbally rate the pain intensity every 10 sec using the numeric pain scale (NPS; "0" meaning 'no pain', "100"- 'worst pain imaginable'). The average pain ratings will be calculated. Temporal summation of heat pain will be defined and calculated as a subtraction of the sixth pain rating (after one minute) from the last pain rating (after two minutes). Hence, a positive value indicates a temporal summation process, and a negative value indicates an adaptation.

The conditioned pain modulation paradigm For assessment of the DNIC efficiency heat stimulation will be delivered using the 3 X 3 cm Peltier based computerized thermal stimulator (TSA, Medoc Ltd, Ramat Yishai, Israel). The baseline temperature will be 32ºC and increase at a rate of 2ºC/sec up to a destination temperature of 46.5ºC and for a duration of 5sec. Patients will verbally report the level of pain intensity using the numeric pain scale (NPS; "0" meaning 'no pain', "100"- 'worst pain imaginable'). This will be considered as 'baseline test pain' (baseline). Then patients will be asked to immerse their dominant hand into a temperature-controlled (10 ºC) water bath (Heto CBN 8-30 Lab equipment, Allerod, Denmark) with a maximum temperature variance of ± 0.5°C, which is continuously stirred by a pump. Following 15 seconds of immersion, while the hand is still in the water bath, a second and third test stimulations will delivered with 15 seconds interval between them, and pain intensity will be recorded again. Two additional heat stimulations will be delivered 15 and 30 seconds subsequent to removal of the hand from the water bath. Upon completion of the session, patients will be instructed to report the intensity of the pain that will be caused by immersing the hand in the water bath (conditioning induced pain intensity). DNIC efficiency will by calculated and define as subtraction of pain ratings of the test stimulus alone from the mean pain ratings of the test stimulus during hand immersion. Thus, negative value indicates greater DNIC efficiency.

Questionnaires SF-MPQ: Short-Form McGill Pain Questionnaire The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors.

Pain related questionnaires Psychological and personality factors known to influence pain perception will be assessed: pain catastrophizing and state and trait anxiety. Assessment will be completed using three questionnaires: (I) The pain catastrophizing scale (PCS), comprised of 13 statements evaluating three dimensions of pain catastrophizing: rumination, magnification and helplessness. Participants will be instructed to rate their agreement with each statement on a scale between 0-4 (0 = "never", 1 = "almost never", 2 = "occasionally", 3 = "almost often", 4 = "often"). The questionnaire score is defined as the sum of all ratings with a high score indicating high pain catastrophizing levels. (II) Spielberger's state-trait anxiety inventory (STAI) that includes two sections each evaluating two distinct features of anxiety: state and trait anxiety. Each section constructed of 20 sentences describing emotional states. Participants will be instructed to rate their emotions about each sentence on a scale between 1-4 (1 = "not at all", 2 = "slightly", 3 = "moderately" 4 = "highly"). The questionnaires score is defined as a sum of all ratings after inverting several specific items, when a high score indicates high levels of state/trait anxiety.

Oswestry Low Back Pain Disability Questionnaire The purpose of the Oswestry Low Back Pain Disability Questionnaire is to assess pain-related disability in persons with low back pain. The questionnaire consists of 10 items addressing different aspects of function. Each item is scored from 0 to 5, with higher values representing greater disability. The total score is multiplied by 2 and expressed as a percentage.

DN4 The DN4 questionnaire consists of 10 items. The first 7 items are related to pain characteristics and sensations and the remaining 3 items are related to the examination. For each item, a score of ''1'' is given if the answer is ''yes'' and a score of ''0'' is given if it is ''no.'' The patient is defined to have neuropathic pain if the sum of all 10 items is calculated to be 4 or more.

Levels of proinflammatory factors in blood and disc tissue Proinflammatory cytokines (IL-1b, IL-6, IL-8, IL-17, TNF-a, INF-g) will be assessed in blood and disc tissue samples obtained at the time of surgery using ProcartaPlex Multiplex Immunoassay and real-time polymerase chain reaction (PCR). All assessments, coding and tissue storage will be held in the Pathology Laboratory at Rambam healthcare campus.

Tissue culture results To minimize the risk of contamination, the surgeon will perform all processing and culturing procedures intraoperatively, and under stringent, sterile, operating theater conditions. During surgery, immediately following intervertebral disc removal, the surgeon will dissect the disc material into 4 proximately equal pieces. PCR method will be used for detection and identification of several bacterial strains from dissected intra-vertebral discs. All assessments, coding and tissue storage will be held in the Microbiology Laboratory at Rambam healthcare campus.

MRI scans of enrolled patients, which are performed regardless to this study protocol, will be evaluated for area and size of the disc protrusion.

Motor examination will be performed using the American Spinal Injury Association (ASIA) score of neurologic assessment. This score will be tested on five muscles in the affected side of the body.

Muscle strength is graded as:

* 0 Total paralysis
* 1 - Palpable or visible contraction
* 2 - Active movement, full range of motion, gravity eliminated
* 3 - Active movement, full range of motion, against gravity
* 4 - Active movement, full range of motion, against gravity and provides some resistance
* 5 - Active movement, full range of motion, against gravity and provides normal resistance [Muscle able to exert, in examiner's judgement, sufficient resistance to be considered normal if identifiable inhibiting factors were not present]
* NT - not testable. Patient unable to reliably exert effort or muscle unavailable for testing due to factors such as immobilization, pain on effort or contracture.

Study procedure All patients scheduled for lumbar spine surgery due to discogenic low back pain and/or sciatica, will be screened by the principal investigator for presence of inclusion/exclusion criteria. Their baseline neurological function before surgery will be assessed and recorded for recruitment into one of the three study groups. MRI scans will be assessed for the calculation of disc protrusion size. Experimental sensory and pain assessments and questionnaires will be performed at list 24 hours before surgery. Blood sample for pro-inflammatory mediator will be obtained at the same time as the experimental sensory and pain tests. Pre-operative pain and MPQ will be assessed pre-operatively (back and leg pain separately), and again on day 30 after surgery. Blood tests for ESR, CRP will be drawn before surgery, during the surgery, and on 30 after surgery. During surgery, intervertebral disc material will be harvested and divided into 4 specimens for culture and inflammatory mediator analysis. Repeat neurological assessment will be performed 30 after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18
2. Capable of understanding the purpose and instructions of the study and signing an informed consent.

Exclusion Criteria:

1) Patients suffering for disc degeneration / herniation or spinal stenosis, scheduled to undergo lumbar spinal surgery for decompression and/or fusion (discectomy, laminectomy, foraminotomy, fusion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 adult subjects suffering from radicular pain duo to disc degeneration / herniation or spinal stenosis will be recruited from the orthopedic clinic at the Rambam Health Care Campus.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Microbial culture and cytokines levels assessed from inter-vertebral disc samples | two years
  Number of positive microbial culture and pro-inflammatory cytokines levels assessed by real-time PCR from intervertebral disc samples

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided